CLINICAL TRIAL: NCT04377724
Title: Longitudinal Serological Study on the Spread and Course of COVID-19 Infections
Brief Title: Spread and Course of COVID-19 Infections
Acronym: CoV-ETH
Status: Completed | Type: Observational
Sponsor: Goldhahn Jörg (Other)
Responsible Party: Sponsor-Investigator, Goldhahn Jörg, Deputy director of the Institute for Translational Medicine, ETH Zurich
Organization: ETH Zurich (Other)
Other Study IDs: 20-05
Record Dates: First submitted 2020-05-05; First posted 2020-05-06 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Covid-19; Virus Disease
MeSH Terms: conditions — COVID-19; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CTG tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ETH cohort: employees or students at ETH Zurich, Switzerland

SUMMARY:
The overall goal is to study the immune response to SARS-CoV-2 infection over the period of one year in the blood of a representative cohort of ETH students/employees.

ELIGIBILITY:
Inclusion Criteria:

* ETH employee or ETH student and their family members living in the same household at the start of the study
* Between 18 and 64 years of age at the start of the study
* Signed informed consent

Exclusion Criteria:

* Age over 64 years at the start of the study
* In quarantine or self-confinement at the start of the study
* Active COVID-19 infection at the start of the study:

  * Diagnosed with a laboratory test
  * Suspected based on typical symptoms such as fever (>38°C), acute pulmonary ex-acerbation or sudden loss of gustatory taste
* The following medical condition

  * With continuous steroid therapy/ chemotherapy/immunsuppressive therapy
  * In treatment for cancer
  * With severe autoimmune disease

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The cohort consists of initially healthy volunteers, all employees or students of ETH. Inclusion into the longitudinal study will be carried out in strict response to the STOP safety concept of the Safety, Security, Health and Environment administrative department of ETH.
Sampling Method: Probability Sample
Enrollment: 2910 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
seroprevalence as well as the titer of serum antibodies (IgM, IgG and IgA) targeting SARS-CoV-2 antigens | 12 months

SECONDARY OUTCOMES:
the property of peripheral blood mononuclear cells before and after an infection with SARS-CoV-2 as opposed to other pathogens | 12 months
the property of IgM and IgA antibody titers against the nucleocapsid protein of SARS-CoV-2 in symptomatic as well as asymptomatic COVID-19 infections over the course of time following an infection | 12 months
the immune response to common-cold (corona)virus and influenza virus infections in patients with COVID-19 infections | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Goldhahn, MD, Study Chair — ETH Zurich; Susanne Ulbrich, Prof. Dr., Study Director — ETH Zurich; Markus Stoffel, Prof. Dr., Study Director — ETH Zurich
Locations (1):
- ETH, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No